CLINICAL TRIAL: NCT06305078
Title: Open-Label Trial of Personalized Medication Experiments to Inform Decisions About Future Attention-Deficit/Hyperactivity Disorder (ADHD) Medication Use
Brief Title: Personalized Attention-Deficit/Hyperactivity Disorder (ADHD) Medication Experiment Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-0528
Record Dates: First submitted 2024-02-13; First posted 2024-03-12 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Open Label Trial
Masking Description: None (open-label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All will choose one of five medication experiment options to complete.
  Interventions: Other: Personalized ADHD Medication Experiment

INTERVENTIONS:
Other: Personalized ADHD Medication Experiment — All parent/adolescent dyads will select and complete a medication experiment.

SUMMARY:
The primary goal of the project is to test personalized medication experiments to inform decisions about future medication use. Our central hypothesis is that our intervention will lead to within subject increases in adolescent involvement in decision making and decreases in uncertainty about future medication use. The investigators view this open label trial as a pilot study to test the feasibility, acceptability, and preliminary efficacy of the medication experiment intervention and therefore warrants further testing in a future larger trial.

DETAILED DESCRIPTION:
The investigators will conduct a pilot, single-arm, open-label trial of the medication experiment intervention among 30 adolescents and parents experiencing uncertainty about continued medicine use. Because the medication experiment intervention is not clinically relevant for adolescents taking a non-stimulant ADHD medication, they will be excluded. At the time of enrollment, families will complete baseline measures electronically and schedule an in-person visit. The investigators will verify the medication prescribed and the number of days covered with medicine in the past year using dispensing data. During the visit, parents and adolescents will choose one of five medication experiments to complete together and track the effects for the desired amount of time.

1. Make no changes. Track current state: continue to take medication as it is currently prescribed.
2. Take medication on non-school days. Track effects: If not currently taking medication on non-school days, start taking medication on those days and track the effects.
3. Stop taking medication on non-school days. Track effects. If currently taking medication on non-school days, stop taking medication on those days and track the effects.
4. Do a formal trial off of medication. Take current medication as currently prescribed for 2 weeks while tracking, then stop taking medication for 2-4 weeks while continuing to track.
5. Change dose or change medication. Consider a different medication or different dose of current medication in consultation with study doctor. Track the effects.

Once dyads have completed the medication experiment, they will complete a follow-up study visit to review the results from the experiment, discuss feasibility of the software, and complete end of study measures.

ELIGIBILITY:
Inclusion Criteria: Participants for the study must meet all of the following criteria:

1. Consent: A parent or legal guardian must provide written informed consent
2. Assent: Adolescents must provide written assent to participate in the study
3. Ages 11-15
4. Treated for ADHD by pediatrician
5. First prescribed ADHD medicine more than one year prior to enrollment
6. Filled at least one prescription for a stimulant medication in the past year
7. Uncertainty about continued ADHD medication use
8. Only one child per household can participate in the study. For families who have more than one child who is potentially eligible, they may decide which of their children would be the best fit for the study.

Exclusion Criteria: Exclusion Criteria: Participants will be excluded from the study if they meet any of the following criteria:

1. Do not have reliable access to the internet at their home or another location.
2. Will not permit their child to access the internet for study related activities.
3. Are not able or willing to send or receive text messages.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Decision-Making Involvement Scale | The investigators will reference the Decision-Making Involvement interview guide to collect this measure at study visit 1 and the stand-alone version 4-12 weeks later at study visit 2.
  A 30-item scale to measure adolescent involvement in a decision. The five subscales are: "Child Seek" (child asks for an opinion or information from parent), "Child Express" (child expresses an opinion or information to parent), "Parent Seek" (parent expresses advice or opinion to child), "Parent Express" (parent expresses advice or opinion to child), and "Joint/Options" (negotiation or brainstorming between parent and child).
Decisional Conflict Scale (DCS) | Collected at study visit 1 and 4-12 weeks later at study visit 2.
  The DCS has an initial question to ascertain the option that has been selected. Options presented will be: continue [medication regimen from experiment], resume previous medication/dosage, conduct another experiment, return to pediatrician to adjust dosage or change medication, other [write in]. The DCS then has 16 questions that are divided into five subscales: informed subscale, values clarity subscale, support subscale, uncertainty subscale, and an effective decision subscale. The total DCS scores are calculated by summing item scores and then converting the scores to a 0-100 scale, where 0 implies no decisional conflict and 100 implies extremely high decisional conflict. Scores <25, 25 to 37.5, >37.5 indicate low, moderate and high decisional conflict, respectively. Scores 25 and higher reflect clinically significant decision conflict.
Behavioral Intention Questions | Collected at study visit 1 and 4-12 weeks later at study visit 2.
  Questions that will assess the adolescent and parent intention to take/give ADHD medicine regularly will be measured using the standard measure of intention from the Unified Theory of Behavior Change. Responses are on a 7-point scale from strongly agree (+3) to strongly disagree (-3) that assess intention to take medicine for ADHD on weekdays, weekends, and school vacations.
System Usability Scale | Collected at study visit 2 (which is 4-12 weeks after study visit 1).
  A validated 10-item unidimensional scale with response options on a 5-point agreement scale which results in a score from 0 to 100, with higher scores indicating greater usability.
Implementation of Decision | 3 months after study visit 2 (which is 4-12 weeks after study visit 1).
  The investigators will obtain pharmacy dispensing records to ascertain whether the dyad's joint decision was implemented. If medication was continued, the investigators will calculate the percentage of days covered.

CONTACTS AND LOCATIONS:
Overall Officials: William Brinkman, MD, MEd, MSc, Principal Investigator — Cincinnati Children's
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT06305078/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT06305078/ICF_001.pdf